CLINICAL TRIAL: NCT06873776
Title: Stimulation-assisted Arm and Leg Cycling for Accelerated Recovery From Spinal Cord Injury
Brief Title: Arm and Leg Cycling for Accelerated SCI Recovery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: University of Alberta (Other)
Responsible Party: Principal Investigator, Jose Pons, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: STU00223113
Record Dates: First submitted 2025-03-07; First posted 2025-03-13 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Spinal Cord Injury
Keywords: Spinal cord injury; Rehabilitation; Cycling; Functional electrical stimulation; transcutaneous spinal cord stimulation; Neuroplasticity
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- A&L_tSCS group (Experimental): This paradigm combines A&L_FES with transcutaneous spinal cord stimulation (tSCS)applied with cathodic electrodes at the C3-C4 and C6-C7 spinous processes and anodic electrodes at the iliac crests. The stimulation intensity is set to trigger a spinal evoked potential, ensuring a strong but tolerable sensation at the cathode sites without evoking direct motor responses in the arm or leg EMG.
  Interventions: Device: A&L cycling
- A&L_FES group (Sham Comparator): This paradigm uses a commercially available motorized ergometer that link the arms & legs mechanically to support voluntary arm and leg cycling and provide reciprocal movements that resemble those during walking. FES is used to assist the the voluntary leg movements, which also enhances proprioceptive feedback. Specifically, functional electrical stimulation (FES) is applied to the major muscles of both legs-including the quadriceps, hamstrings, and gluteus maximus-using pairs of surface electrodes. For sham transcutaneous spinal cord stimulation (tSCS), electrodes will be placed but no tSCS current will be delivered.
  Interventions: Device: A&L cycling
- BWSTT group (Active Comparator): This is the control intervention. Participants will first be assisted by physical therapists/trainers to wear any necessary lower extremity braces along with a padded walking harness. They will then be helped onto the treadmill, either from a wheelchair via a ramp or by walking with physical assistance. Once on the treadmill, they will be clipped into the body weight support system, assisted to a standing position, and provided with the appropriate level of body weight support to facilitate successful stepping.
  Interventions: Device: Body weight supported treadmill training (BWSTT)

INTERVENTIONS:
Device: A&L cycling — Participants will complete simultaneous arms and legs cycling for 60min of active cycling. Targeted exercise intensity is 70-85% of the age-predicted maximum heart rate. Cycling resistance will be modified for continuous challenge. A target speed 10% above the highest speed at which each study participant is able to cycle voluntarily without motor, FES, or tSCS assistance will be selected during the first session and maintained throughout all training sessions. Once a participant can complete 60 minutes of continuous cycling at a specific resistance for two consecutive training sessions, the resistance will be increased to the next setting level at the mid-point of the subsequent session. Upon completion of each session, the physical therapists/researcher will complete skin checks to ensure no adverse effects have occurred. Heart rate, blood pressure, and oxygen saturation will be recorded. Participants will complete 3 training sessions per week for 12 weeks.
  Arms: A&L_FES group; A&L_tSCS group
Device: Body weight supported treadmill training (BWSTT) — The physical therapists/researchers will assist the patient with donning any necessary lower extremity braces and a padded walking harness. The patient will be assisted onto the treadmill via a ramp while seated in a wheelchair or by ambulation with physical assistance, clipped into the body weight support system, assisted to stand, and provided the appropriate amount of body weight support to allow for successful stepping for 60 minutes of active walking. During BWSTT, physical therapists/trainers will adjust treadmill speed or incline and the degree of body weight support to challenge participants. Participants will be instructed to exercise with a targeted intensity of 70-85% of the age-predicted maximum heart rate. Upon completion of each session, the harness will be doffed with skin checks to ensure no adverse effects have occurred. Heart rate, blood pressure, and oxygen saturation will be recorded. Participants will complete 3 training sessions per week for 12 weeks.
  Arms: BWSTT group

SUMMARY:
The purpose of this study is to examine interventions with paradigms involving upper and lower extremity cycling (A&L cycling) with A&L cycling with functional electrical stimulation (FES) (A&L_FES group), A&L cycling with FES and transcutaneous Spinal Cord Stimulation (A&L_tSCS group), and control Body Weight Supported Treadmill Training (BWSTT) to potentially restore functional abilities (i.e., walking) in individuals with an incomplete spinal cord injury. The researchers hypothesize there will be improved walking function following these interventional groups.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) occurs at an annual rate of 50-60 per million in North America. Paralysis is also accompanied by drastic changes in independence and quality of life. SCI occurs mostly among younger individuals, half in people 16-30 years of age. Two-thirds of all SCIs are incomplete (iSCI), with some preserved neural connections relaying information to and from the brain. People with iSCI benefit most from improvements in walking. In addition to increasing independence, walking helps persons with iSCI remain active, with a variety of beneficial health-related outcomes. Therapy that can significantly increase sensorimotor function to these individuals living with iSCI for multiple decades would be hugely significant.

Currently, the most common strategies for restoring walking after an iSCI are manually intensive, including over ground walking with weight and balance support provided by multiple therapists, or with the use of expensive robotic support with controversial outcomes. Thus, the overarching goal of this proposal is to investigate if a non-specific gait rehabilitation paradigm based on motor-assisted arms and legs cycling, motor-assisted arms and legs cycling with functional electrical stimulation (FES) to the main muscles of the legs (A&L_FES group), or motor-assisted arms and legs cycling with FES to the main muscles of the legs and transcutaneous spinal cord stimulation (tSCS) at the cervical level (A&L_tSCS group) in AIS C and D iSCI individuals generalizes to improvements in walking that outperform conventional gait specific training, e.g., body-weight supported treadmill training (BWSTT; control group) (clinical assessments). The researchers will also investigate biomechanical and motor coordination changes and adaptations tied to these functional improvements (biomechanical assessments), and the neural mechanisms that explain functional improvements and their retention over time (neurophysiological assessments).

In the clinical assessments the researchers will investigate the clinically-relevant gait improvements afforded by the cycling intervention by measuring the walking gains with a battery of standard clinical tests focused on motor function, sensation, balance and spasticity. In the biomechanical assessments the researchers will focus on studying the detailed biomechanical basis for the gait improvements by using motion tracking, force plates, and EMG measurement to monitor the kinematics and kinetics of gait, and neuromuscular coordination. In the neurophysiological assessments the researchers will investigate the neuroplastic mechanisms underlying the gait improvements by conducting a battery of physiological tests to detect changes in the strength of descending and ascending spinal pathways.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic or non-traumatic SCI T11 and above (upper motorneuron lesion)
* Incomplete paraplegia or tetraplegia (Classified as AIS C or D)
* Age range 18-75 years old, inclusive
* At least 1 year post- injury
* Independent ambulator (with normal assistive devices or bracing) for at least 10 meters (30 feet)
* Walking speed <0.8 m/s (2.62 ft/s) (or per researcher discretion)
* Bilateral arm strength to arm cycle at least 15 minutes without assistance (or per researcher discretion)
* No concurrent or planned surgeries, significant medical treatments, or therapy during the study period
* Able to understand and speak English

Exclusion Criteria:

* SCI T12 and below (or lacking upper motorneuron injury)
* Complete paraplegia or tetraplegia (classified as AIS A)
* AIS B incomplete paraplegia or tetraplegia
* Presence of progressive neurologic disease
* Unable to give informed consent to participate in the study
* Significant other disease (ex: cardiological or heart disease, renal, hepatic, malignant tumors, mental or psychiatric disorders) that would prevent participants from fullym engaging in study procedures
* Weight over 160 kg (352 lbs)
* TMS contraindications

  * Epilepsy, seizure disorder, or any other type of seizure history
  * Medications that increase the risk of seizures
  * Metal or metal fragments in the head (plates, screws, etc.)
  * Surgical clips in the head or previous neurosurgery
  * Implants in the head (ex: cochlear implants)
  * Non-prescribed drug or marijuana use
  * Depression, antidepressant medications, or antipsychotic medications
* FES and tSCS contraindications

  * Active Deep Vein Thrombosis (blood clot)
  * Active infection in the legs
  * Open wounds, rashes, or infection at the electrode sites
  * Cancer or recently radiated tissue
  * Cardiac pacemakers or neurostimulators
  * Hypersensitivity to or inability to tolerate electrical stimulation
  * Lower motor neuron injury or peripheral nerve injury in the legs that would prevent the muscles from responding to electrical stimulation
* Pregnancy
* Prisoners

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender
Enrollment: 40 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2032-03 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
Change in 10-meter walking test (10MWT) | Changes across baseline, after 3 weeks of training, after 6 weeks of training, after 9 weeks of training, after 12 weeks of training, and 6 months after completing training.
  The 10-meter walking test (10MWT) is a physical function test measuring the total time to ambulate 10 meters in order to calculate walking speed in meters per second. A shorter time indicates a better walking speed.

SECONDARY OUTCOMES:
Change in 6-minute walking test (6MWT) | Changes across baseline, after 3 weeks of training, after 6 weeks of training, after 9 weeks of training, after 12 weeks of training, and 6 months after completing training.
  The 6-minute walking test (6MWT) is a physical function test measuring the total distance walked in a span of six minutes will be assessed. A longer distance indicates a better walking distance.
Change in balance with the Berg balance scale (BBS) | Changes across baseline, after 6 weeks of training, after 12 weeks of training, and 6 months after completing training.
  Change in static and dynamic sitting and standing balance will be assessed using the Berg balance scale (BBS). Items are scored from zero to four. A higher score indicates better balance and decreased fall risk.
Change in walking ability with the WISCI | Changes across baseline, after 6 weeks of training, after 12 weeks of training, and 6 months after completing training.
  The Walking Index for Spinal Cord Injury (WISCI) assesses the ability of a person to walk after spinal cord injury. It consists of a rank ordering at the impairment level from most severe (0) to least severe (20) based on the amount of physical assistance required and use of assistive devices and/or braces while walking a 10-meter distance. A higher score indicates better walking ability.
Change in Modified Ashworth Scale (MAS) | Changes across baseline, after 6 weeks of training, after 12 weeks of training, and 6 months after completing training.
  The Modified Ashworth Scale (MAS) is a physical function test measuring spasticity on a 6-point ordinal scale. A score of 0 on the scale indicates no increase in tone while a score of 4 indicates rigidity. Tone is scored by passively moving the individual's limb and assessing the amount of resistance to movement felt by the examiner. A lower score is a better outcome.
Change in step length | Changes across baseline, after 6 weeks of training, after 12 weeks of training, and 6 months after completing training.
  Step length is the distance between the point of initial contact of one foot and the point of initial contact of the opposite foot. Typically a longer step length is a better outcome, ideally with equal measurements between left and right limbs.
Change in step time | Changes across baseline, after 6 weeks of training, after 12 weeks of training, and 6 months after completing training.
  Step time is the amount of time that passes between the point of initial contact of one foot and the initial contact of the opposite foot. Typically a shorter step time is a better outcome, ideally with equal measurements between left and right limbs.
Change in double support time | Changes across baseline, after 6 weeks of training, after 12 weeks of training, and 6 months after completing training.
  Double support time is the amount of time that passes during which both feet are simultaneously in contact with the ground in a gait cycle. Typically a shorter double support time is a better outcome.
Change in range of motion (ROM) | Changes across baseline, after 6 weeks of training, after 12 weeks of training, and 6 months after completing training.
  Joint angle and angular velocity will be computed with the anatomical neutral position as frame of reference in the sagittal plane and flexion and extension resulting in positive and negative joint angles, respectively. Range of motion will be calculated as the difference between the maximum and minimum hip, knee, and ankle joint angles. A larger range of motion is a better outcome.
Change in joint-joint cyclogram area | Changes across baseline, after 6 weeks of training, after 12 weeks of training, and 6 months after completing training.
  The area inside joint-joint cyclograms (e.g., hip-knee) will be calculated. A larger cyclogram area is a better outcome.
Change in the number of muscle synergies | Changes across baseline, after 6 weeks of training, after 12 weeks of training, and 6 months after completing training.
  Activation patterns and bipolar EMG signals of the leg muscles (gluteus medius, gluteus maximus, rectus femoris, adductor longus, medial hamstrings, tibialis anterior, and gastrocnemius medialis) and arm muscles (delta anterior, delta posterior, biceps brachii, triceps brachii) will be assessed bilaterally during walking. Muscle synergies will be identified from the EMG signals. A higher number of synergies is a better outcome.
Changes in interlimb (upper-lower limb) modulation | Changes across baseline, after 6 weeks of training, after 12 weeks of training, and 6 months after completing training.
  This will be assessed by measuring changes in the magnitude and pattern of H-reflex suppression in the soleus (ankle extensor) of the leg during arm cycling. Features closer to that of a healthy individual is a better outcome.
Changes in the strength of cortico-spinal connectivity | Changes across baseline, after 6 weeks of training, after 12 weeks of training, and 6 months after completing training.
  This will be measured using TMS of the motor cortex known to produce a motor evoked potential (MEP) in the main muscles of the leg, and peak-to-peak amplitude of the MEP and recruitment curves of MEP amplitude as a function of TMS strength will be calculated and constructed. Recruitment curves closer to that of a healthy individual is a better outcome.
Changes in strength of periphery and somatosensory cortex | Changes across baseline, after 6 weeks of training, after 12 weeks of training, and 6 months after completing training.
  This will be measured using cutaneous electrodes on the arm and leg skin surface and recording the somatosensory evoked potentials (SSEPs) over the primary somatosensory cortex using electroencephalography (EEG) electrodes; peak-to-peak amplitude of the SEP and recruitment curves of SEP amplitude as a function of stimulus strength will be calculated and constructed. Recruitment curves closer to that of a healthy individual is a better outcome.

OTHER OUTCOMES:
Change in motor and sensory scores (ASIA) | Changes across baseline, after 6 weeks of training, after 12 weeks of training, and 6 months after completing training.
  The American Spinal Injury Association Impairment Scale (AISA) is a standardized neurological examination used to assess the sensory and motor levels which were affected by the spinal cord injury. A clinician will assess sensory and strength in both upper and lower extremities to provide both a neurologic level of injury and classification level. The five classification levels, ranging from complete loss of neural function in the affected area (Grade A) to completely normal (Grade E). A score closer to Grade E is a better outcome.
Change in functional gait assessment (FGA) | Changes across baseline, after 6 weeks of training, after 12 weeks of training, and 6 months after completing training.
  The FGA is a 10-item test, scored on a four point ordinal scale. A higher score indicates decreased fall risk and is a better outcome. It measures dynamic balance and postural stability during walking tasks (such as fast walking, backward walking, stepping over an obstacle) in the clinical setting. Patients are allowed to use an assistive device for certain items.

CONTACTS AND LOCATIONS:
Overall Officials: Jose L Pons, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No